CLINICAL TRIAL: NCT01287325
Title: A Multi-centre, Randomized, Double-blind, Placebo-controlled, Crossover Study to Evaluate the Clinical Efficacy, Tolerability and Safety of Two Weeks Treatment With DNK333 100 mg Bid in Patients With COPD and Cough.
Brief Title: Efficacy of DNK333 in Patients With COPD and Cough
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DNK333C2201
Record Dates: First submitted 2011-01-26; First posted 2011-02-01 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Cough; DNK333
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cough | interventions — DNK 333

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- DNK333 (Experimental)
  Interventions: Drug: DNK333 100 mg twice daily
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DNK333 100 mg twice daily
  Arms: DNK333
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy and safety of two weeks treatment of DNK333 in patients with COPD and cough.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate COPD
* Forced expiratory volume in 1 second (FEV1) ≥30% predicted
* FEV1/FVC (forced vital capacity) <70%
* Significant amount of cough and minimal amount of sputum production, both as judged by self reporting

Exclusion criteria:

* Upper or lower airway infection within 4 weeks prior to screening
* COPD exacerbation within 4 weeks prior to screening
* Past history or current diagnosis of congestive heart failure, cirrhosis or hepatic failure
* History of lung cancer or pulmonary resection/thoracic radiotherapy

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-09; Primary Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Self-reported cough | At 2 weeks

SECONDARY OUTCOMES:
Sensitivity to capsaicin challenge | At 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, Zuidlaren, Netherlands
- Novartis Investigative Site, London, United Kingdom